CLINICAL TRIAL: NCT03635047
Title: A Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Doses of AL002 in Healthy Participants and in Participants With Mild to Moderate Alzheimer's Disease
Brief Title: A Phase I Study for Safety and Tolerability of AL002.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AL002-1
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Healthy; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AL002 (Active Comparator): AL002 by intravenous (IV) infusion
  Interventions: Biological: AL002
- Saline Solution (Placebo Comparator): placebo by intravenous (IV) infusion
  Interventions: Other: Saline Solution

INTERVENTIONS:
Biological: AL002 — Single-doses of AL002 in up to 9 dose-escalating cohorts
  Arms: AL002
Other: Saline Solution — Saline solution will be administered as a single infusion for each cohort in a ratio of 6 active and 2 placebo subjects for HV and 10 active and 2 placebo for patients
  Arms: Saline Solution

SUMMARY:
This is a multi-centre, randomized, double-blind, placebo-controlled, dose escalation first in human (FIH) study in healthy adults and in patients with mild to moderate Alzheimer's disease. The study is designed to systematically assess the safety (including immunogenicity) and tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of AL002.

DETAILED DESCRIPTION:
The study will be conducted in 2 phases:

In the single ascending dose (SAD) phase up to approximately 56 healthy adult participants will be sequentially enrolled into up to approximately 9 cohorts In the multiple-dose (MD) phase, approximately 32 patients with mild to moderate Alzheimer's disease will be enrolled in three cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Total body weight between 50 and 120 kg, inclusive.
2. Clinical laboratory evaluations (including chemistry panel fasted [fasted at least 8 hours], complete blood count (CBC), and urine analysis) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator. A count of the segmented neutrophils and bands should be performed when results from the white blood cells (WBCs) are not within the reference range.
3. Negative test for selected drugs of abuse at screening (does not include alcohol) and at admission (testing at admission does include alcohol breath test). A positive result may be verified by re-testing (up to one false positive result permitted) and may be followed up at the discretion of the Investigator.
4. Females must be non-pregnant and non-lactating, and either surgically sterile
5. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), laboratory tests, and vital signs.

For MD cohort

1. Ages 50-85 years, inclusive.
2. The participant should be capable of completing assessments alone, per local guidelines.
3. Availability of a person ("study partner") who, in the Investigator's judgment, has frequent and sufficient contact with the participant and is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits, which require partner input for scale completion, and signs the necessary consent form, per local guidelines.
4. Clinical diagnosis of probable Alzheimer's disease dementia based on National Institute on Aging Alzheimer's Association criteria.

Exclusion Criteria:

1. Pregnant or lactating, or intending to become pregnant within 16 weeks after last dose of study drug.
2. Participation in a clinical trial within 30 days before randomization; use of any experimental oral therapy within 30 days or 5 half-lives prior to Day 1, whichever is greater; or use of any biologic therapy within 12 weeks or 5 half-lives prior to Day 1, whichever is greater. Participants who have received an experimental therapy that has no half-life, like a vaccine, should have completed that therapy at least 12 weeks prior to Day 1. Participants who have received an experimental vaccine against a central nervous system (CNS) target, such as beta-amyloid or tau, are not eligible for this study.
3. Any non-experimental vaccine within 2 weeks of randomization, until 2 weeks after the last dose. It is advised that prospective participants receive their annual influenza vaccine as early as possible in advance of the flu season, and then wait 2 weeks prior to randomization. It is permitted to receive the annual influenza vaccine during the screening period.
4. Surgery or hospitalization during the 4 weeks prior to screening.
5. Planned procedure or surgery during the study.
6. Systemically, clinically significantly immunocompromised patients, owing to continuing effects of immune suppressing medication.
7. Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
8. Past history of seizures, with the exception of childhood febrile seizures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of AL002 measured by number of subjects with adverse events and Dose Limiting Adverse Event (DLAEs) | 141 days
  Incidence of adverse events and dose limiting Adverse Events during the DLAE observation period and/or study treatment periods.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AL002 | 85 days
  Serum and CSF concentration of AL002 at specified time points
Maximum plasma concentration (Cmax) for AL002 | 85 days
  Evaluate Cmax for serum and CSF concentration of AL002 at specified time points
Area under the curve concentration (AUC) for AL002 | 85 days
  Evaluate AUC for serum and CSF concentration of AL002 at specified time points

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paul, MD, Study Director — Alector Inc.
Locations (6):
- United States (4):
  - Brain Matters Research, Delray Beach, Florida
  - Compass Research - Orlando, Orlando, Florida
  - Compass Research - The Villages, The Villages, Florida
  - Columbia University, New York, New York
- Nucleus Network Pty Ltd, Melbourne, Australia
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Long H, Simmons A, Mayorga A, Burgess B, Nguyen T, Budda B, Rychkova A, Rhinn H, Tassi I, Ward M, Yeh F, Schwabe T, Paul R, Kenkare-Mitra S, Rosenthal A. Preclinical and first-in-human evaluation of AL002, a novel TREM2 agonistic antibody for Alzheimer's disease. Alzheimers Res Ther. 2024 Oct 23;16(1):235. doi: 10.1186/s13195-024-01599-1. PMID 39444037